CLINICAL TRIAL: NCT00802997
Title: A Double Blind, Randomized, Controlled Trial Assessing Cooled Radiofrequency Denervation as a Treatment fr Sacroiliac Joint Pain Using the Sinergy System
Brief Title: Trial Assessing Cooled Radiofrequency Denervation as a Treatment for Sacroiliac Joint Pain Using the Sinergy System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylis Medical Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SInergy
Record Dates: First submitted 2008-12-04; First posted 2008-12-05 (Estimated); Results first posted 2014-01-01 (Estimated); Last update posted 2014-01-01 (Estimated); Status verified 2013-11

CONDITIONS: Other Acute Pain; Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Treatment with Sinergy system
  Interventions: Device: Sinergy
- 2 (Placebo Comparator): placebo controlled
  Interventions: Device: Placebo sham

INTERVENTIONS:
Device: Sinergy — radiofrequency denervation
  Arms: 1
Device: Placebo sham — sham procedure
  Arms: 2

SUMMARY:
to evaluate the effectiveness of cooled radiotherapy denervation of the sacroiliac region using the sinergy system by comparing a treatment group to a placebo group

ELIGIBILITY:
Inclusion Criteria:

* Predominantly axial pain below L5 vertebrae
* greater than 75%pain relief from 2 seperate lateral branch blocks done on different days
* chronic axial pain lasting longer than 6 months, 3 day average VAS between 4 and 8
* age greater than 18
* failed to acheive adequate improvemnet with comprehensive non-operative treatments, includingbut not limited to: activity alteration, non0steriodal anti-iflammatory, physical and/or manual therap, and flurpscopically guided steriod injections in and around the area of pathology
* all other possible sources oflow back pain have been ruled out, including but not limited to the intervertebral discs, bone fracture.

Exclusion Criteria:

* Beck Depression greater than 20%
* irreversible psychological barriers to recovery
* spinal pathology that may impede recovery such as spins bifida occulta,
* moderate to severe foraminal or central canal stenosis
* systemic infection or localized infection at inducer site
* concomitant cervical or thoracic pain greater than 2/10 on VAS
* uncontrolled or acute disease
* chronic severe condition such as rheumatoid arthritis
* preganancy
* active radicular pain
* immunosuppression
* workers compensation
* allergy to injectants or medications used in procedure
* high narcotis use greater than 30 mg hydrocodone or equivalent
* smokers
* body mass index greater than 29.9

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2008-06; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nileshkumar Patel, MD, Principal Investigator — Coastal Orthopedics & Sports Medicine
Locations (1):
- Coastal Orthopedics & Sports Medicine, Bradenton, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Lateral Branch Neurotomy: The lateral branch neurotomy procedure involved the ablation of the S1-S3 lateral branches and the L5 dorsal ramus using cooled radiofrequency electrodes. The procedure was completed one time within 60 days of enrollment.
- Sham Procedure: The sham procedure was identical to the active treatment procedure but without the delivery of radiofrequency energy. The sham procedure was completed one time within 60 days of enrollment.
Period: Baseline to 3 Months
Arm/Group | Lateral Branch Neurotomy | Sham Procedure
Started | 34 | 17
Completed | 34 | 17
Not Completed | 0 | 0
Period: 3 Months to 6 Months
Arm/Group | Lateral Branch Neurotomy | Sham Procedure
Started | 34 | 0 (Sham subjects unblinded at 3 Months. None continued in sham group.)
Completed | 27 | 0 (Sham subjects unblinded at 3 Months. None continued in sham group.)
Not Completed | 7 | 0
Period: 6 Month to 9 Months
Arm/Group | Lateral Branch Neurotomy | Sham Procedure
Started | 27 | 0 (Sham subjects unblinded at 3 Months. None continued in sham group.)
Completed | 25 | 0 (Sham subjects unblinded at 3 Months. None continued in sham group.)
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lateral Branch Neurotomy | Sham Procedure | Total
Number analyzed (Participants) | 34 | 17 | 51
Age Continuous [Mean (Standard Deviation); unit: years] | 56 (15) | 64 (14) | 59 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 14 | 37
  Male | 11 | 3 | 14
Region of Enrollment [Number; unit: participants]
  United States | 34 | 17 | 51
Sacroiliac Joint Pain Intensity [Mean (Standard Deviation); unit: Units on a scale] — Scale ranges from 0 to 10. A score of 0 represents no pain and a score of 10 represents the highest level of pain.
  Units on a scale | 6.1 (1.3) | 5.8 (1.3) | 6.0 (1.3)

OUTCOME MEASURES:

1. Primary Outcome: Pain Status Change for Sacroiliac Joint Pain Intensity
Description: Scale ranges from 0 to 10. A score of 0 represents no pain and a score of 10 represents the highest level of pain.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lateral Branch Neurotomy | Sham Procedure
Number analyzed (Participants) | 34 | 17
units on a scale | -2.4 (2.7) | -0.8 (2.4)
Statistical Analysis 1: Comparison: Lateral Branch Neurotomy vs Sham Procedure; Test type: Superiority or Other; p = 0.035, t-test, 2 sided

2. Other Pre Specified Outcome: Pain Status Change for Sacroiliac Joint Pain Intensity
Description: Scale ranges from 0 to 10. A score of 0 represents no pain and a score of 10 represents the highest level of pain.
Time Frame: Baseline and 6 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lateral Branch Neurotomy | Sham Procedure
Number analyzed (Participants) | 27 | 0
units on a scale | -2.5 (2.6) |

3. Other Pre Specified Outcome: Pain Status Change for Sacroiliac Joint Pain Intensity
Description: Scale ranges from 0 to 10. A score of 0 represents no pain and a score of 10 represents the highest level of pain.
Time Frame: Baseline and 9 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lateral Branch Neurotomy | Sham Procedure
Number analyzed (Participants) | 25 | 0
units on a scale | -2.7 (2.7) |

ADVERSE EVENTS:
Arm/Group | Lateral Branch Neurotomy | Sham Procedure
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/17
Other Adverse Events (participants affected / at risk) | 0/34 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results communications must be provided to the Sponsor for review 30 days prior to public release. The Sponsor has the right to review materials for the purposes of preserving confidentiality of Sponsor's proprietary information, which may be removed at the Sponsor's request, and for identification of patentable inventions. The Investigator has no obligation to address any additional comments provided during the review and has final control and approval of publication content.